CLINICAL TRIAL: NCT03948087
Title: Comparison of Wound Healing, Edema Level, Knee Range of Motion, Protection Post Falls, Device Application, Time to Prosthetic Fit, and Cost Between Postoperative Soft Dressing and Vacuum Removable Rigid Dressing After Transtibial Amputation
Brief Title: Comparison Between Postoperative Tubular Dressing and a Vacuum Removable Rigid Dressing After Transtibial Amputation
Acronym: EMPAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Covenant Health, Canada (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Trent Duchscherer, Amputee Coordinator Northern Alberta Vascular Center, Covenant Health, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMPAR
Record Dates: First submitted 2019-02-27; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Amputation Stump; Peripheral Vascular Disease With Complications; Edema Leg; Wound Healing Delayed

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an interventional group (vacuum rigid removable dressing) vs a non-interventional group (standard of care control group of soft dressing application).
Who Masked: Outcomes Assessor
Masking Description: Wound assessments will be determined in a blinded capacity by utilizing the Photographic Wound Assessment Tool. Photos of individual study participant's wounds will be taken and then assigned a non-identifying marker prior to being submitted by the wound assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum Removable Rigid Dressing (VRRD) (Experimental): Application of a Vacuum Removable Rigid Dressing (VRRD)
  Interventions: Device: Vacuum Removable Rigid Dressing (VRRD)
- Soft Dressing Control Group (No Intervention): Application of standard of care soft dressing (SD) intra-operatively.

INTERVENTIONS:
Device: Vacuum Removable Rigid Dressing (VRRD) — Intra-operative application of device.
  Other Names: Ossur (TM) Rigid Dressing (ORD)
  Arms: Vacuum Removable Rigid Dressing (VRRD)

SUMMARY:
Comparison of wound healing, edema level, knee range of motion, rate of revision post falls, device application time, time to prosthetic fit, and cost between postoperative soft dressing and a vacuum removable rigid dressing after unilateral transtibial amputation.

DETAILED DESCRIPTION:
The gold standard after transtibial amputation is casting of the residual limb to limit room for post-surgical edema, enable faster wound healing and shorter hospital stays, as well as, reduce time to prosthetic fitting. Casting also reduces the risk of impact damage to the limb. Casting, however, is costly and impractical due to the requirement of a prosthetist available on call for after emergency amputation surgeries and a need for multiple repeat prosthetist visits to cut off and reapply casting after wound healing checks. Thus current practice involves use of a compression elastic tube bandage (like a tensor bandage) applied within 15 minutes after surgery. However this bandage applies pressure to the residual limb, which can increase risk of reduced blood supply to the healing limb especially in vascular compromised patients. Further, this soft bandage does not offer any protection to the residual limb, a fall or severe contusion could lead to a requirement for costly revision surgery. There is evidence that rigid removable dressings can improve wound healing times, protect the limb, prevent contractures and enable earlier prosthetic fitting. This study aims to examine the the differences in wound healing time, changes in limb edema, knee range of motion, limb protection post falls, device application time, time to prosthetic fitting and cost between currently used postoperative soft dressing (SD) and vacuum removable rigid dressing (VRRD) after transtibial amputation.

ELIGIBILITY:
Inclusion Criteria:

1. Transtibial amputation related to peripheral vascular disease with or without diabetes or trauma.

   Justification: The form and function of the ORD device relates solely to transtibial amputees. The device is not useable for any other limb amputation type (e.g. transfemoral, transmetatarsal). The choice of using vascular compromised participants is intentional. Ischemia and necrosis rapidly ensue as a result of vessel occlusion which can easily happen with any external compressive force (e.g. tensor bandaging). The ORD does not apply compressive force to the residual limb.
2. Transtibial amputation that includes myodesis and/or myoplasty.

   Justification: Myoplasty and myodesis are preferred surgical techniques while performing an amputation. They involve the surgical attachment of muscle to muscle (myoplasty) or muscle to bone (myodesis) across the end of the residual limb prior to skin flap closure. This allows increased stability and provides a better interface with a future prosthetic device.
3. Greater than 18 years of age

   Justification: Below the age of 18 informed consent must be obtained by a parent or guardian
4. Patient must be able to speak and understand English in order to provide informed consent. No reliance on translator services will be implemented.
5. Has no major illness where life expectancy is less than 2 years.

Justification: This is the study timeline and co-morbidities that limit participation within this timeframe will introduce confounding factors.

Exclusion Criteria:

1. Severe dementia or insufficient cognition.

   Justification: Inability to provide informed consent to participate in the study.
2. Knee contracture greater than 30 degrees

   Justification: The ORD will not fit a limb with too much flexion at the knee. Wound healing is also affected due to pressure across the end of the residual limb without the use of offloading techniques.
3. Severe peripheral vascular disease involving the contralateral lower limb

   Justification: Having severe peripheral vascular disease to the contralateral limb may affect the secondary outcome measures due to the need for further medical or surgical intervention.
4. Inability to speak, read, or understand English.

   Justification: For a patient to participate in the study informed consent must be obtained. There is a high probability that there would be too much variability among translators (family member or institutional) to ensure consistent informed consent.
5. Neurological condition or medical disorder that could affect rehabilitation.

Justification: Rehabilitation post transtibial amputation is critical to overall functional outcomes as well as study outcomes. If a patient has difficulty with participation in rehabilitation then this will be a confounding factor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Change in Stump Wound Healing | Day 3,7,14,30,48
  The Photographic Wound Assessment Tool (PWAT) will be used in a blinded fashion to evaluate the level of change in wound healing of the transtibial amputation primary closure. The PWAT incorporates type and amount of necrotic tissue, wound edge definition, surrounding skin color, epithelialization, and granulation of tissue. A score of 0/24 on the PWAT indicates complete wound closure.

SECONDARY OUTCOMES:
Evaluation of Change in Level of Limb Edema | Day 3,7,14,30,48
  Circumferential measurements will be taken at two levels of the residual stump. Centimeters measured circumferentially at 5 cm from the distal end and around the knee at the center of the patella
Evaluation of Change in Knee Range of Motion | Day 3,7,14,30,48
  Degrees measured via goniometry into knee flexion and extension for both active and passive range of motion.
Rate of Revision Post Falls | Until prosthetic limb fit, on average 2 months.
  Falls sustained by study participants will be recorded. Whether a follow-up revision surgery was necessary will also be recorded.
Total Amount of Time to Apply, Change, Clean and Alter the Dressings | Until discharge from acute care, on average 2 weeks.
  Time log in minutes recorded by staff in real time providing care to study participants.
Length of time Until the Residual Limb is Ready for Prosthetic Fitting | Through study completion, on average 2 months.
  Time log in days beginning post operative day 1 until the study participant is fit with a definitive prosthetic limb.
Total Length of Stay in Acute and Sub-acute Care Facilities | Through study completion, on average 3 weeks.
  A time log in days of how long a given study participant is admitted to an acute or sub-acute care facility.

CONTACTS AND LOCATIONS:
Overall Officials: Trent I Duchscherer, MSc, Principal Investigator — Amputee Coordinator Northern Alberta Vascular Center; Gerrit B Winkelaar, MD, Study Director — Divisional Director and Clinical Head of Vascular Surgery for the Edmonton zone

IPD SHARING:
Plan to Share IPD: No